CLINICAL TRIAL: NCT04014413
Title: Safety and Efficacy of Fecal Microbiota Transplantation: A Pilot Study
Brief Title: Safety and Efficacy of Fecal Microbiota Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMT-Pilot
Record Dates: First submitted 2019-06-21; First posted 2019-07-10 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Crohn Disease; Ulcerative Colitis; Celiac Disease; Irritable Bowel Syndrome; Functional Dysphonia; Constipation; Clostridium Difficile Infection; Diabetes Mellitus; Obesity; Multidrug -Resistant Infection; Hepatic Encephalopathy; Multiple Sclerosis; Pseudo-Obstruction; Carbapenem-Resistant Enterobacteriaceae Infection; Vancomycin Resistant Enterococci Infection; Multiple Organ Dysfunction Syndrome; Dysbiotic Bowel Syndrome; MRSA Enteritis; Pseudomembranous Enterocolitis; Alopecia; Autism; Graft-versus-host Disease; Idiopathic Thrombocytopenic Purpura; Atopy or Allergy; Liver Disease; Alcohol Dependence; Psoriatic Arthropathy
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Celiac Disease; Irritable Bowel Syndrome; Constipation; Clostridium Infections; Diabetes Mellitus; Obesity; Hepatic Encephalopathy; Multiple Sclerosis; Multiple Organ Failure; Enterocolitis, Pseudomembranous; Alopecia; Autistic Disorder; Graft vs Host Disease; Purpura, Thrombocytopenic, Idiopathic; Hypersensitivity; Liver Diseases; Alcoholism; Arthritis, Psoriatic | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (25):
- Crohn's disease (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Ulcerative colitis (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Celiac disease (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Irritable bowel syndrome (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Functional dyspepsia (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Constipation (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Metabolic disease (diabetes mellitus or obesity) (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Multidrug-resistant infection (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Hepatic encephalopathy (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Multiple sclerosis (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Pseudo-obstruction (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- CRE infection (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- VRE infection (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Multiple organ dysfunction (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Dysbiotic bowel syndrome (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- MRSA enteritis (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Pseudomembranous enteritis (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Alopecia (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Autism (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Graft-versus-host disease (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Idiopathic thrombocytopenic purpura (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Atopy or allergy (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Liver disease (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Alcohol dependence (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Antibiotic-associated diarrhea (Experimental): Fecal Microbiota Transplant will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation

INTERVENTIONS:
Procedure: Fecal Microbiota Transplantation — Fecal microbiota transplantation

SUMMARY:
The gut microbiota is critical to health and functions with a level of complexity comparable to that of an organ system. Dysbiosis, or alterations of this gut microbiota ecology, have been implicated in a number of disease states. Fecal microbiota transplantation (FMT), defined as infusion of feces from healthy donors to affected subjects, is a method to restore a balanced gut microbiota and has attracted great interest in recent years due to its efficacy and ease of use. FMT is now recommended as the most effective therapy for CDI not responding to standard therapies.

Recent studies have suggested that dysbiosis is associated with a variety of disorders, and that FMT could be a useful treatment. Randomized controlled trial has been conducted in a number of disorders and shown positive results, including alcoholic hepatitis, Crohn's disease (CD), ulcerative colitis (UC), pouchitis, irritable bowel syndrome (IBS), hepatic encephalopathy and metabolic syndrome. Case series/reports and pilot studies has shown positive results in other disorders including Celiac disease, functional dyspepsia, constipation, metabolic syndrome such as diabetes mellitus, multidrug-resistant, hepatic encephalopathy, multiple sclerosis, pseudo-obstruction, carbapenem-resistant Enterobacteriaceae (CRE) or Vancomycin-resistant Enterococci (VRE) infection, radiation-induced toxicity, multiple organ dysfunction, dysbiotic bowel syndrome, MRSA enteritis, Pseudomembranous enteritis, idiopathic thrombocytopenic purpura (ITP), and atopy.

Despite FMT appears to be relatively safe and efficacious in treating a wide range of disease, its safety and efficacy in a usual clinical setting is unknown. More data is required to confirm safety and efficacy of FMT. Therefore, the investigators aim to conduct a pilot study to investigate the efficacy and safety of FMT in a variety of dysbiosis-associated disorder.

ELIGIBILITY:
Inclusion Criteria:

Confirmed diagnosis of any of the following diseases:

* Crohn's disease
* Ulcerative colitis
* Celiac disease
* Irritable bowel syndrome
* Functional dyspepsia
* Constipation
* Antibiotic-associated diarrhea or any antibiotic- associated complications/symptoms
* Metabolic syndrome such as diabetes mellitus and obesity
* Multidrug-resistant infection
* Hepatic encephalopathy
* Multiple sclerosis
* Pseudo-obstruction
* Carbapenem-resistant Enterobacteriaceae (CRE) or Vancomycin-resistant Enterococci (VRE) infection
* Multiple organ dysfunction
* Dysbiotic bowel syndrome
* MRSA enteritis
* Pseudomembranous enteritis
* Alopecia, autism
* Graft-versus-host disease
* Idiopathic thrombocytopenic purpura (ITP)
* Atopy or allergy
* Liver disease such as Nonalcoholic fatty liver disease (NAFLD) and Nonalcoholic steatohepatitis (NASH)
* Alcohol dependence
* Psoriatic arthropathy that has suboptimal control of disease despite standard treatment.

Exclusion Criteria:

* Known contraindication to all FMT infusion method such as nasoduodenal tube insertion, oesophago-gastro-duodenoscopy (OGD), enteroscopy, colonoscopy and enema
* Any conditions that may render the efficacy of FMT or at the discretion of the investigators
* Current pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2030-10-31 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
The efficacy of FMT in treating dysbiosis-associated disorder will be assessed by number of patients who have improvement in clinical symptoms (depends on each disease as stated in outcome) | 1 year

SECONDARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | 1 year

OTHER OUTCOMES:
Any improvement or deterioration or recurrence of the underlying condition by clinical judgement of doctors | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Siew Ng, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brandt LJ. American Journal of Gastroenterology Lecture: Intestinal microbiota and the role of fecal microbiota transplant (FMT) in treatment of C. difficile infection. Am J Gastroenterol. 2013 Feb;108(2):177-85. doi: 10.1038/ajg.2012.450. Epub 2013 Jan 15. PMID 23318479
- [Background] Philips CA, Pande A, Shasthry SM, Jamwal KD, Khillan V, Chandel SS, Kumar G, Sharma MK, Maiwall R, Jindal A, Choudhary A, Hussain MS, Sharma S, Sarin SK. Healthy Donor Fecal Microbiota Transplantation in Steroid-Ineligible Severe Alcoholic Hepatitis: A Pilot Study. Clin Gastroenterol Hepatol. 2017 Apr;15(4):600-602. doi: 10.1016/j.cgh.2016.10.029. Epub 2016 Nov 2. No abstract available. PMID 27816755
- [Background] Yang Z, Wang X, Bu C. Fecal microbiota transplant for Crohn's disease: a prospective, randomized study in chinese population. United european gastroenterology journal. Conference: 25th united european gastroenterology week, UEG 2017. Spain. Volume 5, 2017:A112-a113
- [Background] Paramsothy S, Kamm MA, Kaakoush NO, Walsh AJ, van den Bogaerde J, Samuel D, Leong RWL, Connor S, Ng W, Paramsothy R, Xuan W, Lin E, Mitchell HM, Borody TJ. Multidonor intensive faecal microbiota transplantation for active ulcerative colitis: a randomised placebo-controlled trial. Lancet. 2017 Mar 25;389(10075):1218-1228. doi: 10.1016/S0140-6736(17)30182-4. Epub 2017 Feb 15. PMID 28214091
- [Background] Rossen NG, Fuentes S, van der Spek MJ, Tijssen JG, Hartman JH, Duflou A, Lowenberg M, van den Brink GR, Mathus-Vliegen EM, de Vos WM, Zoetendal EG, D'Haens GR, Ponsioen CY. Findings From a Randomized Controlled Trial of Fecal Transplantation for Patients With Ulcerative Colitis. Gastroenterology. 2015 Jul;149(1):110-118.e4. doi: 10.1053/j.gastro.2015.03.045. Epub 2015 Mar 30. PMID 25836986
- [Background] Moayyedi P, Surette MG, Kim PT, Libertucci J, Wolfe M, Onischi C, Armstrong D, Marshall JK, Kassam Z, Reinisch W, Lee CH. Fecal Microbiota Transplantation Induces Remission in Patients With Active Ulcerative Colitis in a Randomized Controlled Trial. Gastroenterology. 2015 Jul;149(1):102-109.e6. doi: 10.1053/j.gastro.2015.04.001. Epub 2015 Apr 7. PMID 25857665
- [Background] Costello SP, Waters O, Bryant RV, et al. Short duration, low intensity, pooled fecal microbiota transplantation induces remission in patients with mildmoderately active ulcerative colitis: A randomised controlled trial. Gastroenterology 2017;152 (5 Supplement 1):S198-S199
- [Background] Kirk KF, Kousgaard SJ, Nielsen HL, et al. Faecal transplant for the treatment of chronic pouchitis-A randomised, placebo-controlled, clinical trial. Colorectal Disease 2017;19 (Supplement 2):143
- [Background] Johnsen PH, Hilpusch F, Cavanagh JP, et al. Fecal transplantation in Irritable Bowel Syndrome (IBS): An RCT. Neurogastroenterology and Motility 2017;29 (Supplement 2):135.
- [Background] Holster S, Repsilber D, Brummer RJ, et al. Faecal microbiota transfer in irritable bowel syndrome-clinical outcomes of a randomised placebo-controlled trial. United European Gastroenterology Journal 2017;5 (5 Supplement 1):A155-A156.
- [Background] Holster S, Brummer RJ, Repsilber D, et al. Fecal microbiota transplantation in irritable bowel syndrome and a randomized placebo-controlled trial. Gastroenterology 2017;152 (5 Supplement 1):S101-S102.
- [Background] Holger Johnsen P, Mazzawi T, El-Salhy M, et al. Effect of faecal microbiota transplantation on the enteroendocrine cells of the colon in patients with Irritable Bowel Syndrome (IBS): Double blinded-placebo controlled study. Neurogastroenterology and Motility 2017;29 (Supplement 2):71.
- [Background] Bajaj JS, Kassam Z, Fagan A, et al. Fecal microbiota transplant using a precision medicine approach is safe, Associated with lower hospitalization risk and improved cognitive function in recurrent hepatic encephalopathy. Journal of Hepatology 2017;66:S49-S49.
- [Background] Mullish BH, McDonald JAK, Thursz MR, Marchesi JR. Fecal microbiota transplant from a rational stool donor improves hepatic encephalopathy: A randomized clinical trial. Hepatology. 2017 Oct;66(4):1354-1355. doi: 10.1002/hep.29369. Epub 2017 Aug 26. No abstract available. PMID 28714089